CLINICAL TRIAL: NCT05447169
Title: Parallel Controlled Study of Epstein-Barr Virus Antibody and Epstein-Barr Virus DNA for Nasopharyngeal Carcinoma Screening in the High-risk Population
Brief Title: Epstein-Barr Virus Antibody and Epstein-Barr Virus DNA for Nasopharyngeal Carcinoma Screening
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); Hunan Cancer Hospital (Other); The Third Affiliated Hospital of Nanchang University (Other); First People's Hospital of Foshan (Other); Yuebei People's Hospital (Other); Xiangya Hospital of Central South University (Other); Changsha Central Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Other Study IDs: SYSUCC-CMY-2022-screen
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma Screen; EBV DNA; EBV antibody
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal brushing and peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High risk population of nasopharyngeal carcinoma: first-degree relatives of nasopharyngeal carcinoma patients, aged 30-62 male
  Interventions: Diagnostic Test: EBV antibodies test; Diagnostic Test: EBV DNA test

INTERVENTIONS:
Diagnostic Test: EBV antibodies test — ELISA test of VCA-IgA，EBNA1-IgA，EA-IgA， Zta-IgA ，Rta-IgG and BNLF 2b in nasopharyngeal brushing and plasma
Diagnostic Test: EBV DNA test — quantitative polymerase chain reaction, CRISPR-associated protein 12a and target sequencing of EBV DNA in nasopharyngeal brushing and plasma

SUMMARY:
The investigators intend to compare Epstein-Barr virus antibody and Epstein-Barr virus DNA screening efficacy in first-degree relatives of nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
The investigators intend to test Epstein-Barr virus antibodies (Viral Capsid Antigen-immunoglobulin A， Epstein-Barr nuclear antigen 1-immunoglobulin A， early antigen-immunoglobulin A， Zta-immunoglobulin A， Rta-immunoglobulin G, Bnlf 2b) by ELISA and Epstein-Barr virus DNA by quantitative polymerase chain reaction, target sequencing and CRISPR-associated protein 12a in nasopharyngeal brushing and plasma of the same population at high-risk of nasopharyngeal carcinoma so as to determine the best method in nasopharyngeal carcinoma screening.

ELIGIBILITY:
Inclusion Criteria:

* residents in Southern China
* 30-62 years old
* male
* a first-degree relative of at least one nasopharyngeal carcinoma patient
* no medical record of nasopharyngeal carcinoma
* Eastern Cooperative Oncology Group score of 0-2
* be able to comprehend, sign, and date the written informed consent document to participate in the study

Exclusion Criteria:

* history of nasopharyngeal carcinoma
* heavy cardiovascular, liver or kidney disease
* on systemic steroid or immunosuppressant treatment or active autoimmune disease

Ages: 30 Years to 62 Years | Sex: Male
Age Groups: Adult
Study Population: Residences in Southern China
Sampling Method: Non-Probability Sample
Enrollment: 11625 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
positive predictive value | 3 years
  the ratio of subjects truly diagnosed as nasopharyngeal carcinoma to all those who had positive test results
negative predictive value | 3 years
  the ratio of subjects truly diagnosed as negative (do not have nasopharyngeal carcinoma) to all those who had negative test results

SECONDARY OUTCOMES:
sensitivity | 3 years
  the percentage of subjects who test positive to those who have nasopharyngeal carcinoma
specificity | 3 years
  the percentage of subjects who test negative to those who do not have nasopharyngeal carcinoma
early diagnose rate | 3 years
  the ratio of patients with stage I and stage II disease to all those who have nasopharyngeal carcinoma
cost-effectiveness | 3 years
  the cost of detecting one nasopharyngeal carcinoma case

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China